CLINICAL TRIAL: NCT01490047
Title: Phase I Trial of Intravenous Recombinant Human TNF-α and Liposomal Doxorubicin in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: Single Dose of Intravenous rhTNF-α and Liposomal Doxorubicin in Patients With Advanced Solid Tumors or Lymphomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2011-001
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Solid Tumors; Lymphomas
MeSH Terms: conditions — Lymphoma | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- rhTNF-α 25 µg/m² + Caelyx 40 mg/m² (Experimental): Cohort 2: rhTNF-α 25 µg/m² + Caelyx 40 mg/m²
  Interventions: Drug: Recombinant human TNF-α; Drug: Liposomal doxorubicin; Drug: Caelyx
- rhTNF-α 50 µg/m² + Caelyx 40 mg/m² (Experimental): Cohort 3: rhTNF-α 50 µg/m² + Caelyx 40 mg/m²
  Interventions: Drug: Recombinant human TNF-α; Drug: Liposomal doxorubicin; Drug: Caelyx
- rhTNF-α 100 µg/m² + Caelyx 40 mg/m² (Experimental): Cohort 4: rhTNF-α 100 µg/m² + Caelyx 40 mg/m²
  Interventions: Drug: Recombinant human TNF-α; Drug: Liposomal doxorubicin; Drug: Caelyx
- rhTNF-α 150 µg/m² + Caelyx 40 mg/m² (Experimental): Cohort 5: rhTNF-α 150 µg/m² + Caelyx 40 mg/m²
  Interventions: Drug: Recombinant human TNF-α; Drug: Liposomal doxorubicin; Drug: Caelyx
- rhTNF-α 200 µg/m² + Caelyx 40 mg/m² (Experimental): Cohort 6: rhTNF-α 200 µg/m² + Caelyx 40 mg/m²
  Interventions: Drug: Recombinant human TNF-α; Drug: Liposomal doxorubicin; Drug: Caelyx
- rhTNF-α 250 µg/m² + Caelyx 40 mg/m² (Experimental): Cohort 7: rhTNF-α 250 µg/m² + Caelyx 40 mg/m²
  Interventions: Drug: Recombinant human TNF-α; Drug: Caelyx
- rhTNF-α 25 µg/m² + Caelyx 30 mg/m² (Experimental): Cohort 1 rhTNF-α 25 µg/m² + Caelyx 30 mg/m²
  Interventions: Drug: Recombinant human TNF-α; Drug: Liposomal doxorubicin; Drug: Caelyx

INTERVENTIONS:
Drug: Recombinant human TNF-α — Infusion will be done over 60 minutes, preferably via central venous catheter. Will immediately follow the infusion of Liposomal doxorubicin.
  Other Names: Beromun
Drug: Liposomal doxorubicin — Infusion over 60 minutes
  Other Names: Caelyx
  Arms: rhTNF-α 100 µg/m² + Caelyx 40 mg/m²; rhTNF-α 150 µg/m² + Caelyx 40 mg/m²; rhTNF-α 200 µg/m² + Caelyx 40 mg/m²; rhTNF-α 25 µg/m² + Caelyx 30 mg/m²; rhTNF-α 25 µg/m² + Caelyx 40 mg/m²; rhTNF-α 50 µg/m² + Caelyx 40 mg/m²
Drug: Caelyx — Administration of Caelyx® will be done first, as infusion in 250 ml D5W, followed immediately by infusion of rhTNF-α.
  Other Names: liposomal doxorubicin
Drug: Recombinant human TNF-α — Recombinant human TNF-α (Beromun) will be diluted in 250 mL of normal saline with albumin (2 mg/mL) to prevent adherence of the protein to the delivery apparatus. Infusion will be done over 60 minutes, preferably via central venous catheter, including PICC lines.
  Other Names: Beromun

SUMMARY:
Assess the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of recombinant human tumor necrosis factor-α (rhTNF-α) when given as a single dose intravenously and in combination with liposomal doxorubicin in human subjects

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a diagnosed solid tumor malignancy or lymphoma indicated for Caelyx treatment.
* Patient is refractory to all lines of standard therapy including biologics, chemo or other therapies, or at least one line of therapy in those patients for whom no standard treatment exists.
* Patient has measurable disease (defined as at least one lesion whose longest diameter can be accurately measured as >1 cm).
* At least 2 weeks has elapsed since the completion of the last cycle of chemotherapy and/or major surgery and the patient is fully recovered from this previous therapy or surgery and any post-surgical complications.
* The patient has a normal cardiac ejection fraction on MUGA or Echocardiogram.
* ECOG performance status of 2 or less.
* Patient is at least 18 years of age.
* Patient is capable of giving informed consent.
* Patient of childbearing potential is using adequate birth control measures (e.g., abstinence, barrier method with spermicide; intrauterine device, implantable or injectable contraceptives or surgical sterilization) for the duration of the study and will continue to use such precautions for 12 months after receiving treatment.

Exclusion Criteria:

* Positive pregnancy test or known pregnancy.
* Participation in any other clinical trial
* Known hypersensitivity to the active substance or to any of the excipients (Albumin).
* Patients exposed to greater than 450 mg/m2 of doxorubicin or Caelyx.
* Patient has a creatinine > 1.5 x the upper limit of normal, chronic renal failure requiring hemodialysis or peritoneal dialysis.
* Platelet count equal to or less than 50,000/mm3, Hemoglobin less than 9.0 g/dL, or an ANC less than 1,000 /mm3.
* Patient has a Sa02 of less than 93% on room air.
* Patient with detectable ascites or portosystemic hypertension or cirrhosis.
* Patient with bilirubin > 2.0, AST or ALT above 2.5X the upper limit of normal, an alkaline phosphatase above 2.5X the upper limit of normal.
* Hypercalcaemia > 12 mg/dl (2.99 mmol/l).
* Patients with contraindications to the use of vasopressor substances.
* Patient has presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to screening) or bone marrow transplant.
* Patient has a history of a significant medical illness deemed by the principal investigator or sub-investigators as unsuitable for the trial, for example: Significant cardiovascular disease, e.g. congestive heart failure (New York Heart Association Class II, III or IV), severe angina pectoris, cardiac arrhythmias, myocardial infarction within a 3 month period prior to treatment, venous thrombosis, occlusive peripheral arterial disease, recent pulmonary embolism. Severe pulmonary dysfunction. A recent history of, or active peptic ulcer. Severe ascites. Known hypotension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of a single dose of intravenous recombinant human tumor necrosis factor-α plus liposomal doxorubicin | Up to 22 days
  MTD is the dose level below the one that produces 2 or more Dose-Limiting Toxicities
Dose Limiting Toxicity (DLT) of a single dose of intravenous recombinant human tumor necrosis factor-α plus liposomal doxorubicin | up to 22 days
  Toxicity Criteria will be those listed in NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  Any grade 3 cytokine release syndrome/acute infusion reaction or allergic and toxicity Grade 3 and above will be considered a DLT except:
  * Grade 3 toxicities that recover to grade 1 or less within 48 hours after standard supportive treatment.
  * Grade 4 neutropenia that recovers within 14 days.
  * Grade 4 thrombocytopenia that recovers within 14 days.
  * Grade 4 anemia that recovers within 14 days.

SECONDARY OUTCOMES:
Overall tumor response using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | 4 weeks
Caelyx/doxorubicin plasma levels | 0, 24, 48 and 192 hours post-dose
  Caelyx/doxorubicin plasma levels will be measured at 0, 24, 48 and 192 hours post-dose by fluorimetry (excitation at 470nm, emission 590 nm) after liposomes have been disrupted in 70% ethanol, 0.3 N HCl

CONTACTS AND LOCATIONS:
Overall Officials: Elke Jäger, MD, Principal Investigator — Krankenhaus Nordwest, Frankfurt, Germany
Locations (1):
- Krankenhaus Nordwest, Frankfurt, Germany